CLINICAL TRIAL: NCT03950115
Title: Effects and Prognostic Factors of Intensive Pulse Light Treatment for Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, tae-young chung, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-04-066
Record Dates: First submitted 2019-04-22; First posted 2019-05-15 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): IPL therapy will be performed with the M22® (Lumenis, Dreieich, Germany). IPL treatment is going to be administered to the skin below the lower eyelid. Before treatment, the eyes will be protected with opaque goggles. Ultrasound gel is going to be applied to the patient's face from tragus to tragus including the nose in order to conduct the light, help to spread the energy evenly, and provide a degree of protection. The intensity of the IPL treatment will range from 9.8J/cm2 to 13J/cm2 according to Fitzpatrick Skin Type Grading.
  Interventions: Device: Intense Pulsed Light (IPL)

INTERVENTIONS:
Device: Intense Pulsed Light (IPL) — IPL therapy will be performed with the M22® (Lumenis, Dreieich, Germany). IPL treatment is going to be administered to the skin below the lower eyelid. Before treatment, the eyes will be protected with opaque goggles. Ultrasound gel is going to be applied to the patient's face from tragus to tragus including the nose in order to conduct the light, help to spread the energy evenly, and provide a degree of protection. The intensity of the IPL treatment will range from 9.8J/cm2 to 13J/cm2 according to Fitzpatrick Skin Type Grading.
  Other Names: Meibomian gland expression

SUMMARY:
The investigators are going to Investigate the comparative efficacy of intense pulsed light therapy alone with that of intense pulsed light plus meibomian gland expression for meibomian gland dysfunction.

DETAILED DESCRIPTION:
Enrolled patients are going to be randomly assigned to two groups. All of the patients will undergo four treatment sessions in total, which are two weeks apart. Group 1 will undergo two sessions of intense pulsed light therapy with meibomian gland expression, as well as two sessions of intense pulsed light alone. Group 2 will receive two sessions of intense pulsed light therapy alone, and two sessions of intense pulsed light therapy with meibomian gland expression. The following parameters will be measured at baseline, 2 weeks after the second treatment session, and 2 weeks after the fourth treatment session: tearfilm break-up time, Oxford grade for corneal staining, meibomian gland expressibility, meibum quality, and ocular surface disease index.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of meibomian gland dysfunction

Exclusion Criteria:

* Medical conditions in which IPL is contraindicated (pregnancy, breastfeeding, lupus, and any major uncontrolled health problem).
* Contact lens wearer
* Previous ocular surgery
* Previous thermal treatment for dry eye disease (e.g. LipiFlow)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline tearfilm break-up time at 2 weeks after the last treatment session | Baseline and 2 weeks after the last treatment session
Change from baseline Oxford grade for corneal staining at 2 weeks after the last treatment session | Baseline and 2 weeks after the last treatment session
  Oxford grade for staining was assessed on a scale of 0 to 5. It was scaled according to the degree of corneal staining as follow: 0 (absent), 1 (minimal), 2 (mild), 3 (moderate), 4 (marked), and 5 (severe)
Change from baseline meibomian gland expressibility score at 2 weeks after the last treatment session | Baseline and 2 weeks after the last treatment session
  The meibomian gland expressibility was assessed on a scale of 0 to 3 in ﬁve glands on the central lower lid. It was scaled according to the number of glands expressible, as follows: 0 (all glands), 1 (three to four glands), 2 (one to two glands) and 3 (no glands)
Change from baseline meibum quality score at 2 weeks after the last treatment session | Baseline and 2 weeks after the last treatment session
  The meibum quality score were divided into the following four degrees: 0 (clear), 1 (cloudy), 2 (granular), and 3 (toothpaste)
Change from baseline ocular surface disease index at 2 weeks after the last treatment session | Baseline and 2 weeks after the last treatment session
  The ocular surface diseases index score range from 0 to 100 based on the result of standardized ocular surface disease index questionnaire. Higher value represent worse subjective symptom.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No